CLINICAL TRIAL: NCT03906396
Title: Investigating the Feasibility of Exergame on Sleep and Emotion Among University Students
Brief Title: Exergame on Sleep and Emotion Among Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Principal Investigator, Farahiyah Wan Yunus, Principal Investigator, National University of Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NN-2018-167
Record Dates: First submitted 2019-04-03; First posted 2019-04-08 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Depression; Sleep; Anxiety; Stress
Keywords: xbox kinect; gaming technology; stress; anxiety; depression; randomised control trial; sleep quality; intervention
MeSH Terms: conditions — Depression; Anxiety Disorders; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Intervention group: Using the Xbox 360 Kinect Control Group: No intervention, continue with daily routine
Who Masked: Outcomes Assessor
Masking Description: i) A number of assessors from occupational therapy students will be recruited. This is to allow for randomization possibility on assessment responsibility.
  1. Pre-evaluation is conducted randomly by accident by an independent assessor with an occupational therapy background without knowing which participant in which group. There is no specific client on specific assessor.
  2. The post-evaluation is conducted randomly by accident by an independent assessor with an occupational therapy background. There is no specific client on specific assessor.
  ii) Information among participants is kept confidential and blinding from each other. No cross-over is allowed to reduce bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): A session 30 minutes of exercise game activities using the Xbox 360 Kinect will be performed by each participant for 6 weeks, 3 times per week. Games use for the activity are Sports Kinect and Sports Kinect 2. The activity can be performed in solo or in pairs with another participant. The game activity will be played only at the site chosen for this study.
  Interventions: Device: Xbox 360 Kinect
- Control Group (No Intervention): No standard activity is provided for the participants. The participants will continue with their normal daily life activities.

INTERVENTIONS:
Device: Xbox 360 Kinect — A session 30 minutes of exercise game activities using the Xbox 360 Kinect will be performed by each participant. Games uses for the activity are Sports Kinect and Sports Kinect 2. Xbox 360 Kinect - the players themselves become the ''game controller'' via their body movements and gestures, Kinect-enabled game titles lend themselves comfortably to the class of exercise games.
  Arms: Intervention Group

SUMMARY:
This study aims to investigate the feasibility and the potential efficacy of using Xbox 360 Kinect game among healthcare undergraduate students. Thirty-six participants will be recruited and randomly allocated into the intervention and control group. The session will be 30 minutes per session for three times per week. Two outcome measures will be used at pre and post intervention.

DETAILED DESCRIPTION:
Sleep deprivation and emotional problems such as stress, anxiety and depression commonly occur in university students. Exercise is beneficial to ameliorate those problems however university students are not serious to uptake physical activity. Commercially available exergame such as Xbox 360 Kinect is one of the alternatives. This study aims to investigate the feasibility and the potential efficacy of using Xbox 360 Kinect game among healthcare undergraduate students. A pilot two-armed parallel randomized controlled trial was implemented. A total of 36 undergraduate students was recruited and randomly allocated into the intervention group (playing Xbox 360 Kinect) or the control group (continue with normal daily routine). The intervention group received 30 minutes of Xbox Kinect activity, three times per week for six weeks. Information on psychology (DASS-21) and sleep (FOSQ-30) status were collected at pre- and post-experiment. The researcher-developed feasibility questionnaire was given to the participants in the intervention group at post-experiment. Repeated-measures ANOVA analysis was used to investigate within-between group comparison and significant value was set at p≤0.05. The analysis found potential improvement on sleep (p=0.039) and psychological health (p=0.002-0.067). The intervention protocol is feasible and highly accepted by the participants. Required optimum amount of dosage, sample size and used of outcome measures are suggested from the findings. This pilot and feasibility study support the use of Xbox 360 Kinect games in practice and to be implemented for future research.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate healthcare students
* Able to read and understand English version questionnaire
* Having BMI <25

Exclusion Criteria:

* Person with condition (i.e. asthma, heart problem) that prevent from participating in active physical activities.
* Known history of mental health issues
* Visually impaired students iv. Postgraduate students

Ages: 19 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-04-07 (Actual)

PRIMARY OUTCOMES:
Depression, Anxiety and Stress Scales Questionnaire (DASS-21) | 1 week
  The Depression, Anxiety and Stress Scale -21 Items (DASS-21) is a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress. Each of the three DASS-21 scales contains 7 items, divided into subscales with similar content. Scores for depression, anxiety and stress are calculated by summing the scores for the relevant items. Scoring for each scale is from 0 to 3 (Never:0; Sometimes:1; Often:2; Almost Always:3). Overall score is summed to indicate if the person has depression, anxiety or stress. For depression total score indicators (Normal:0-4; Mild:5-6; Moderate:7-10; Severe:11-13; Extremely Severe:14+). For anxiety total score indicators (Normal: 0-3; Mild:4-5; Moderate:6-7; Severe: 8-9; Extremely Severe: 10+). For stress total score indicators (Normal:0-7; Mild: 8-9; Moderate: 10-12; Severe: 13-16; Extremely Severe: 17+)
Functional Outcome of Sleep Questionnaire (FOSQ-30) | 1 week
  Consisting of 30 questions related to the effects of fatigue on daily activities, the instrument was designed to evaluate the respondent's quality of life as it relates to disorders of excessive sleepiness. In 30 items, the FOSQ then assesses difficulty, due to sleepiness, in performing activities of daily living and recreational activities, which are categorized into the following 5 subscales: 1) activity level (9 items), 2) vigilance (7 items), 3) intimacy and sexual relationships (4 items), 4) general productivity (8 items), and 5) social outcomes (2 items). Scoring is from 0-4 (0: I don't do this activity for other reasons; 1: Yes, Extremely Difficult; 2: Yes, Moderate Difficulty; 3: Yes, Little Difficulty: 4: No Difficulty. The potential range of scores for the Total Score is 5 -20. Lower Score indicates more difficulty performing everyday activities when tired or sleepy, while higher score indicates less difficulty performing everyday activities when tired or sleepy.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Hibatullah Romli, PhD, Principal Investigator — Universiti Putra Malaysia
Locations (1):
- Kolej Tun Syed Nasir, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No
Study protocol can be shared with other researchers